CLINICAL TRIAL: NCT00038727
Title: Diabetes Prevention Program Outcomes Study
Acronym: DPPOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Aging (NIA) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); National Eye Institute (NEI) (NIH); National Center for Research Resources (NCRR) (NIH); Office of Research on Women's Health (ORWH) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); American Diabetes Association (Other); Indian Health Service (IHS) (U.S. Federal Agency); General Clinical Research Program (Unknown); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DPPOS; U01DK048489 (NIH); NCT00353314 (obsolete NCT alias)
Record Dates: First submitted 2002-06-04; First posted 2002-06-05 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus; Cancer; CVD
Keywords: DPP; IGT; Prediabetes; Type 2 diabetes; Macrovascular disease; Microvascular disease; Lifestyle; Metformin; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms; Prediabetic State; Diabetes Mellitus, Type 2; Obesity | interventions — Metformin

STUDY DESIGN:
Masking Description: Open label phase for metformin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 Original Lifestyle (Active Comparator): randomized to unmasked Intensive Lifestyle during the DPP and offered Intensive Lifestyle Group Session, DPPOS Group Lifestyle plus DPPOS Boost Lifestyle sessions in DPPOS Phase 1 and 2
  Interventions: Behavioral: DPPOS Group Lifestyle; Behavioral: DPPOS Boost Lifestyle; Behavioral: Intensive Lifestyle Group Session
- 2 Original Metformin (Active Comparator): randomized to the masked metformin treatment group during DPP and continued open label in DPPOS. Participants were also offered Intensive Lifestyle Group Session, DPPOS Group Lifestyle in DPPOS Phase 1 and 2.
  Interventions: Behavioral: DPPOS Group Lifestyle; Drug: Metformin; Behavioral: Intensive Lifestyle Group Session
- 3 Original Placebo (Placebo Comparator): randomized to masked placebo during DPP and offered Intensive Lifestyle Group Session, DPPOS Group Lifestyle in DPPOS Phase 1 and 2
  Interventions: Behavioral: DPPOS Group Lifestyle; Behavioral: Intensive Lifestyle Group Session

INTERVENTIONS:
Behavioral: DPPOS Group Lifestyle — Quarterly group lifestyle sessions
Drug: Metformin — Administered as 850mg twice per day, masked in DPP and open label in DPPOS
  Other Names: Glucophage
  Arms: 2 Original Metformin
Behavioral: DPPOS Boost Lifestyle — In addition to quarterly group, 2 additional classes per year and an annual 15 minute check-up.
  Arms: 1 Original Lifestyle
Behavioral: Intensive Lifestyle Group Session — 16 session curriculum in group format. In DPP delivered to ILS as individual sessions
  Other Names: Intensive lifestyle session (ILS)

SUMMARY:
The Diabetes Prevention Program (DPP) was a multi-center trial examining the ability of an intensive lifestyle or metformin to prevent or delay the development of diabetes in a high risk population due to the presence of impaired glucose tolerance (IGT, 2 hour glucose of 140-199 mg/dl). The DPP has ended early demonstrating that lifestyle reduced diabetes onset by 58% and metformin reduced diabetes onset by 31%.

DPPOS (2002-2013) is designed to take advantage of the scientifically and clinically valuable DPP participants. This group of participants is nearly 50% minority and represents the largest at risk population ever studied. Clinically important research questions remain that focus on 1) durability of the prior DPP intervention, 2) determination of the clinical course of precisely known new onset diabetes, in particular regarding microvascular disease, CVD risk factors and atherosclerosis, 3) close examination of these topics in men vs women and in minority populations.

The major aims of DPPOS-3 (2014-2025) take advantage of the long-term randomized exposure of the study cohort to metformin and the aging of the DPPOS cohort. The metformin exposure and high degree of study retention and adherence (~85% of the DPPOS cohort continues to attend annual and mid-year visits) allows DPPOS-3 to examine the long-term effects of metformin on cardiovascular disease (CVD) and cancer outcomes, outcomes of great clinical interest and import.

DETAILED DESCRIPTION:
The current DPPOS Executive Summary and protocol, as well as DPPOS protocol and lifestyle manuals and publications are available at: http://www.dppos.org

ELIGIBILITY:
Participation as a volunteer in the Diabetes Prevention Program (DPP).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2779 (Actual)
Dates: Start 2002-09; Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Nathan, MD, Study Chair — Massachusetts General Hospital; Marinella Temprosa, PhD, Principal Investigator — George Washington University Biostatistics Center; Barbara Linder, MD, PhD, Study Director — NIDDK Project Scientist; Kishore Gadde, MD, Principal Investigator — Pennington Biomedical Research Center; David Ehrmann, MD, Principal Investigator — University of Chicago; Kevin Furlong, MD, Principal Investigator — Jefferson Medical College of Thomas Jefferson University; Kathleen Jablonski, PhD, Principal Investigator — George Washington University Biostatistics Center; Ronald B Goldberg, MD, Principal Investigator — University of Miami; Helen P Hazuda, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Dana Dabelea, MD, PhD, Principal Investigator — University of Colorado, Denver; Medha Munshi, MD, Principal Investigator — Joslin Diabetes Center; Steven Kahn, MB, ChB, Principal Investigator — University of Washington; Samuel Dagogo-Jack, MD, MB, Principal Investigator — University of Tennessee; Mark Molitch, MD, Principal Investigator — Northwestern University; Happy Araneta, PhD,MPH, Principal Investigator — University of California, San Diego; F. Xavier Pi-Sunyer, MD, Principal Investigator — Columbia University; Kieren J Mather, MD, Principal Investigator — Indiana University; Michelle Magee, MD, Principal Investigator — Medstar Health Research Institute; Karol E Watson, MD, Principal Investigator — University of California, Los Angeles; Angela Brown, MD, Principal Investigator — Washington University School of Medicine; Sherita Hill Golden, MD, MHS, Principal Investigator — Johns Hopkins School of Medicine; David S Schade, MD, Principal Investigator — The University of New Mexico; Jill Crandall, MD, Principal Investigator — Albert Einstein College of Medicine; Elizabeth Venditti, PhD, Principal Investigator — University of Pittsburgh; Marjerie Mau, MD, Principal Investigator — University of Hawaii; William Knowler, MD, Principal Investigator — SW Indian Center, NIDDK; Santica M Marcovina, PhD, Principal Investigator — University of Washington; David M Nathan, MD, Principal Investigator — Massachusetts General Hospital; Christine Lee, MD, Study Director — NIDDK Project Scientist; Sunder Mudaliar, MD, Principal Investigator — University of California, San Diego
Locations (1):
- George Washington University, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Repository
Time Frame: 2002-2025
Access Criteria: Instructions for access are detailed here: https://repository.niddk.nih.gov/pages/overall_instructions/
URL: https://repository.niddk.nih.gov/studies/dppos/

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Result] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986
- [Result] Diabetes Prevention Program Research Group. Long-term effects of lifestyle intervention or metformin on diabetes development and microvascular complications over 15-year follow-up: the Diabetes Prevention Program Outcomes Study. Lancet Diabetes Endocrinol. 2015 Nov;3(11):866-75. doi: 10.1016/S2213-8587(15)00291-0. Epub 2015 Sep 13. PMID 26377054
- [Derived] Lin PD, Cardenas A, Temprosa M, Botelho JC, Calafat AM, Gold DR, Oken E, Fleisch AF. Associations of Perfluoroalkyl and Polyfluoroalkyl Substances With Cardiovascular Disease Incidence in Adults With Prediabetes: Findings From the Diabetes Prevention Program. J Am Heart Assoc. 2026 Jan 6;15(1):e046298. doi: 10.1161/JAHA.125.046298. Epub 2025 Dec 18. PMID 41413398
- [Derived] Tjaden AH, Goldbaum AA, Edelstein SL, Heckman-Stoddard BM, Reedy J, Herman WH, Hoskin M, Knowler WC, Schlogl M, Temple KA, Venditti EM, Watson K, Temprosa M, Shams-White MM; DPP Research Group. The 2018 World Cancer Research Fund/American Institute for Cancer Research Score and Cancer Risk: results from the diabetes prevention program outcomes study. Am J Clin Nutr. 2025 Sep;122(3):715-723. doi: 10.1016/j.ajcnut.2025.07.011. Epub 2025 Jul 15. PMID 40675492
- [Derived] Knowler WC, Doherty L, Edelstein SL, Bennett PH, Dabelea D, Hoskin M, Kahn SE, Kalyani RR, Kim C, Pi-Sunyer FX, Raghavan S, Shah VO, Temprosa M, Venditti EM, Nathan DM; DPP/DPPOS Research Group. Long-term effects and effect heterogeneity of lifestyle and metformin interventions on type 2 diabetes incidence over 21 years in the US Diabetes Prevention Program randomised clinical trial. Lancet Diabetes Endocrinol. 2025 Jun;13(6):469-481. doi: 10.1016/S2213-8587(25)00022-1. Epub 2025 Apr 28. PMID 40311647
- [Derived] Munshi MN, Venditti EM, Tjaden AH, Knowler WC, Boyko EJ, Middelbeek RJW, Luchsinger JA, Lee CG, Hazuda HP, Salive ME, Edelstein SL, Storer TW. Long-term impact of Diabetes Prevention Program interventions on walking endurance. Front Public Health. 2024 Dec 18;12:1470035. doi: 10.3389/fpubh.2024.1470035. eCollection 2024. PMID 39744353
- [Derived] Gadde KM, Yin X, Goldberg RB, Orchard TJ, Schlogl M, Dabelea D, Ibebuogu UN, Watson KE, Pi-Sunyer FX, Crandall JP, Temprosa M, Luchsinger JA; Diabetes Prevention Program Research Group. Coronary Artery Calcium and Cognitive Decline in the Diabetes Prevention Program Outcomes Study. J Am Heart Assoc. 2023 Nov 7;12(21):e029671. doi: 10.1161/JAHA.123.029671. Epub 2023 Nov 6. PMID 37929764
- [Derived] Molitch ME, Tripputi M, Levey AS, Crandall JP, Dabelea D, Herman WH, Knowler WC, Orchard TJ, Schroeder EB, Srikanthan P, Temprosa M, White NH, Nathan DM; Diabetes Prevention Program Research Group. Electronic address: dppmail@bsc.gwu.edu. Effects of metformin and intensive lifestyle interventions on the incidence of kidney disease in adults in the DPP/DPPOS. J Diabetes Complications. 2023 Sep;37(9):108556. doi: 10.1016/j.jdiacomp.2023.108556. Epub 2023 Jul 25. PMID 37607422
- [Derived] Shams-White MM, Tjaden AH, Edelstein SL, Bassiouni S, Kahle LL, Kim C, Pi-Sunyer X, Temple KA, Venditti EM, Reedy J, Heckman-Stoddard BM; DPP Research Group. The 2018 World Cancer Research Fund (WCRF)/American Institute for Cancer Research (AICR) score and diabetes risk in the Diabetes Prevention Program Outcomes Study (DPPOS). BMC Nutr. 2022 Sep 21;8(1):105. doi: 10.1186/s40795-022-00596-7. PMID 36131333
- [Derived] Goldberg RB, Orchard TJ, Crandall JP, Boyko EJ, Budoff M, Dabelea D, Gadde KM, Knowler WC, Lee CG, Nathan DM, Watson K, Temprosa M; Diabetes Prevention Program Research Group*. Effects of Long-term Metformin and Lifestyle Interventions on Cardiovascular Events in the Diabetes Prevention Program and Its Outcome Study. Circulation. 2022 May 31;145(22):1632-1641. doi: 10.1161/CIRCULATIONAHA.121.056756. Epub 2022 May 23. PMID 35603600
- [Derived] Lee CG, Heckman-Stoddard B, Dabelea D, Gadde KM, Ehrmann D, Ford L, Prorok P, Boyko EJ, Pi-Sunyer X, Wallia A, Knowler WC, Crandall JP, Temprosa M; Diabetes Prevention Program Research Group; Diabetes Prevention Program Research Group:. Effect of Metformin and Lifestyle Interventions on Mortality in the Diabetes Prevention Program and Diabetes Prevention Program Outcomes Study. Diabetes Care. 2021 Dec;44(12):2775-2782. doi: 10.2337/dc21-1046. Epub 2021 Oct 25. PMID 34697033
- [Derived] Varga TV, Liu J, Goldberg RB, Chen G, Dagogo-Jack S, Lorenzo C, Mather KJ, Pi-Sunyer X, Brunak S, Temprosa M; Diabetes Prevention Program Research Group. Predictive utilities of lipid traits, lipoprotein subfractions and other risk factors for incident diabetes: a machine learning approach in the Diabetes Prevention Program. BMJ Open Diabetes Res Care. 2021 Mar;9(1):e001953. doi: 10.1136/bmjdrc-2020-001953. PMID 33789908
- [Derived] Kriska AM, Rockette-Wagner B, Edelstein SL, Bray GA, Delahanty LM, Hoskin MA, Horton ES, Venditti EM, Knowler WC; DPP Research Group. The Impact of Physical Activity on the Prevention of Type 2 Diabetes: Evidence and Lessons Learned From the Diabetes Prevention Program, a Long-Standing Clinical Trial Incorporating Subjective and Objective Activity Measures. Diabetes Care. 2021 Jan;44(1):43-49. doi: 10.2337/dc20-1129. Epub 2020 Nov 10. PMID 33444158
- [Derived] Hazuda HP, Pan Q, Florez H, Luchsinger JA, Crandall JP, Venditti EM, Golden SH, Kriska AM, Bray GA. Association of Intensive Lifestyle and Metformin Interventions With Frailty in the Diabetes Prevention Program Outcomes Study. J Gerontol A Biol Sci Med Sci. 2021 Apr 30;76(5):929-936. doi: 10.1093/gerona/glaa295. PMID 33428709
- [Derived] Kim C, Younes N, Temprosa M, Edelstein S, Goldberg RB, Araneta MG, Wallia A, Brown A, Darwin C, Ibebuogu U, Pi-Sunyer X, Knowler WC. Infertility, Gravidity, and Risk Of Diabetes among High-Risk Women in the Diabetes Prevention Program Outcomes Study. J Clin Endocrinol Metab. 2020 Mar 1;105(3):e358-67. doi: 10.1210/clinem/dgaa013. PMID 31955207
- [Derived] Perreault L, Pan Q, Schroeder EB, Kalyani RR, Bray GA, Dagogo-Jack S, White NH, Goldberg RB, Kahn SE, Knowler WC, Mathioudakis N, Dabelea D; Diabetes Prevention Program Research Group. Regression From Prediabetes to Normal Glucose Regulation and Prevalence of Microvascular Disease in the Diabetes Prevention Program Outcomes Study (DPPOS). Diabetes Care. 2019 Sep;42(9):1809-1815. doi: 10.2337/dc19-0244. Epub 2019 Jul 18. PMID 31320445
- [Derived] Cardenas A, Hivert MF, Gold DR, Hauser R, Kleinman KP, Lin PD, Fleisch AF, Calafat AM, Ye X, Webster TF, Horton ES, Oken E. Associations of Perfluoroalkyl and Polyfluoroalkyl Substances With Incident Diabetes and Microvascular Disease. Diabetes Care. 2019 Sep;42(9):1824-1832. doi: 10.2337/dc18-2254. Epub 2019 Jul 11. PMID 31296647
- [Derived] Apolzan JW, Venditti EM, Edelstein SL, Knowler WC, Dabelea D, Boyko EJ, Pi-Sunyer X, Kalyani RR, Franks PW, Srikanthan P, Gadde KM; Diabetes Prevention Program Research Group. Long-Term Weight Loss With Metformin or Lifestyle Intervention in the Diabetes Prevention Program Outcomes Study. Ann Intern Med. 2019 May 21;170(10):682-690. doi: 10.7326/M18-1605. Epub 2019 Apr 23. PMID 31009939
- [Derived] Diabetes Prevention Program Research Group. Long-term Effects of Metformin on Diabetes Prevention: Identification of Subgroups That Benefited Most in the Diabetes Prevention Program and Diabetes Prevention Program Outcomes Study. Diabetes Care. 2019 Apr;42(4):601-608. doi: 10.2337/dc18-1970. PMID 30877090
- [Derived] Cardenas A, Hauser R, Gold DR, Kleinman KP, Hivert MF, Fleisch AF, Lin PD, Calafat AM, Webster TF, Horton ES, Oken E. Association of Perfluoroalkyl and Polyfluoroalkyl Substances With Adiposity. JAMA Netw Open. 2018 Aug 3;1(4):e181493. doi: 10.1001/jamanetworkopen.2018.1493. PMID 30646133
- [Derived] Kim C, Ricardo AC, Boyko EJ, Christophi CA, Temprosa M, Watson KE, Pi-Sunyer X, Kalyani RR; Diabetes Prevention Program Research Group. Sex Hormones and Measures of Kidney Function in the Diabetes Prevention Program Outcomes Study. J Clin Endocrinol Metab. 2019 Apr 1;104(4):1171-1180. doi: 10.1210/jc.2018-01495. PMID 30398516
- [Derived] DeBoer MD, Filipp SL, Gurka MJ. Use of a Metabolic Syndrome Severity Z Score to Track Risk During Treatment of Prediabetes: An Analysis of the Diabetes Prevention Program. Diabetes Care. 2018 Nov;41(11):2421-2430. doi: 10.2337/dc18-1079. Epub 2018 Oct 1. PMID 30275282
- [Derived] Kim C, Aroda VR, Goldberg RB, Younes N, Edelstein SL, Carrion-Petersen M, Ehrmann DA; Diabetes Prevention Program Outcomes Study Group. Androgens, Irregular Menses, and Risk of Diabetes and Coronary Artery Calcification in the Diabetes Prevention Program. J Clin Endocrinol Metab. 2018 Feb 1;103(2):486-496. doi: 10.1210/jc.2017-01829. PMID 29220533
- [Derived] Crandall JP, Mather K, Rajpathak SN, Goldberg RB, Watson K, Foo S, Ratner R, Barrett-Connor E, Temprosa M. Statin use and risk of developing diabetes: results from the Diabetes Prevention Program. BMJ Open Diabetes Res Care. 2017 Oct 10;5(1):e000438. doi: 10.1136/bmjdrc-2017-000438. eCollection 2017. PMID 29081977
- [Derived] Perreault L, Pan Q, Aroda VR, Barrett-Connor E, Dabelea D, Dagogo-Jack S, Hamman RF, Kahn SE, Mather KJ, Knowler WC; Diabetes Prevention Program Research Group. Exploring residual risk for diabetes and microvascular disease in the Diabetes Prevention Program Outcomes Study (DPPOS). Diabet Med. 2017 Dec;34(12):1747-1755. doi: 10.1111/dme.13453. Epub 2017 Sep 19. PMID 28833481
- [Derived] Aroda VR, Knowler WC, Crandall JP, Perreault L, Edelstein SL, Jeffries SL, Molitch ME, Pi-Sunyer X, Darwin C, Heckman-Stoddard BM, Temprosa M, Kahn SE, Nathan DM; Diabetes Prevention Program Research Group. Metformin for diabetes prevention: insights gained from the Diabetes Prevention Program/Diabetes Prevention Program Outcomes Study. Diabetologia. 2017 Sep;60(9):1601-1611. doi: 10.1007/s00125-017-4361-9. Epub 2017 Aug 2. PMID 28770322
- [Derived] Herman WH. The cost-effectiveness of diabetes prevention: results from the Diabetes Prevention Program and the Diabetes Prevention Program Outcomes Study. Clin Diabetes Endocrinol. 2015 Sep 2;1:9. doi: 10.1186/s40842-015-0009-1. eCollection 2015. PMID 28702228
- [Derived] Kim C, Dabelea D, Kalyani RR, Christophi CA, Bray GA, Pi-Sunyer X, Darwin CH, Yalamanchi S, Barrett-Connor E, Golden SH, Boyko EJ. Changes in Visceral Adiposity, Subcutaneous Adiposity, and Sex Hormones in the Diabetes Prevention Program. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3381-3389. doi: 10.1210/jc.2017-00967. PMID 28651370
- [Derived] Luchsinger JA, Ma Y, Christophi CA, Florez H, Golden SH, Hazuda H, Crandall J, Venditti E, Watson K, Jeffries S, Manly JJ, Pi-Sunyer FX; Diabetes Prevention Program Research Group. Metformin, Lifestyle Intervention, and Cognition in the Diabetes Prevention Program Outcomes Study. Diabetes Care. 2017 Jul;40(7):958-965. doi: 10.2337/dc16-2376. Epub 2017 May 12. PMID 28500216
- [Derived] Goldberg RB, Aroda VR, Bluemke DA, Barrett-Connor E, Budoff M, Crandall JP, Dabelea D, Horton ES, Mather KJ, Orchard TJ, Schade D, Watson K, Temprosa M; Diabetes Prevention Program Research Group. Effect of Long-Term Metformin and Lifestyle in the Diabetes Prevention Program and Its Outcome Study on Coronary Artery Calcium. Circulation. 2017 Jul 4;136(1):52-64. doi: 10.1161/CIRCULATIONAHA.116.025483. Epub 2017 May 5. PMID 28476766
- [Derived] Aroda VR, Edelstein SL, Goldberg RB, Knowler WC, Marcovina SM, Orchard TJ, Bray GA, Schade DS, Temprosa MG, White NH, Crandall JP; Diabetes Prevention Program Research Group. Long-term Metformin Use and Vitamin B12 Deficiency in the Diabetes Prevention Program Outcomes Study. J Clin Endocrinol Metab. 2016 Apr;101(4):1754-61. doi: 10.1210/jc.2015-3754. Epub 2016 Feb 22. PMID 26900641
- [Derived] Marrero DG, Ma Y, de Groot M, Horton ES, Price DW, Barrett-Connor E, Carnethon MR, Knowler WC; Diabetes Prevention Program Research Group. Depressive symptoms, antidepressant medication use, and new onset of diabetes in participants of the diabetes prevention program and the diabetes prevention program outcomes study. Psychosom Med. 2015 Apr;77(3):303-10. doi: 10.1097/PSY.0000000000000156. PMID 25775165
- [Derived] Aroda VR, Christophi CA, Edelstein SL, Zhang P, Herman WH, Barrett-Connor E, Delahanty LM, Montez MG, Ackermann RT, Zhuo X, Knowler WC, Ratner RE; Diabetes Prevention Program Research Group. The effect of lifestyle intervention and metformin on preventing or delaying diabetes among women with and without gestational diabetes: the Diabetes Prevention Program outcomes study 10-year follow-up. J Clin Endocrinol Metab. 2015 Apr;100(4):1646-53. doi: 10.1210/jc.2014-3761. Epub 2015 Feb 23. PMID 25706240
- [Derived] Diabetes Prevention Program Research Group. HbA1c as a predictor of diabetes and as an outcome in the diabetes prevention program: a randomized clinical trial. Diabetes Care. 2015 Jan;38(1):51-8. doi: 10.2337/dc14-0886. Epub 2014 Oct 21. PMID 25336746
- [Derived] Diabetes Prevention Program (DPP) Research Group; Hamman RF, Horton E, Barrett-Connor E, Bray GA, Christophi CA, Crandall J, Florez JC, Fowler S, Goldberg R, Kahn SE, Knowler WC, Lachin JM, Murphy MB, Venditti E. Factors affecting the decline in incidence of diabetes in the Diabetes Prevention Program Outcomes Study (DPPOS). Diabetes. 2015 Mar;64(3):989-98. doi: 10.2337/db14-0333. Epub 2014 Oct 2. PMID 25277389
- [Derived] Dabelea D, Ma Y, Knowler WC, Marcovina S, Saudek CD, Arakaki R, White NH, Kahn SE, Orchard TJ, Goldberg R, Palmer J, Hamman RF; Diabetes Prevention Program Research Group. Diabetes autoantibodies do not predict progression to diabetes in adults: the Diabetes Prevention Program. Diabet Med. 2014 Sep;31(9):1064-8. doi: 10.1111/dme.12437. Epub 2014 Apr 9. PMID 24646311
- [Derived] Marrero D, Pan Q, Barrett-Connor E, de Groot M, Zhang P, Percy C, Florez H, Ackermann R, Montez M, Rubin RR; DPPOS Research Group. Impact of diagnosis of diabetes on health-related quality of life among high risk individuals: the Diabetes Prevention Program outcomes study. Qual Life Res. 2014 Feb;23(1):75-88. doi: 10.1007/s11136-013-0436-3. Epub 2013 May 26. PMID 23709097
- [Derived] Price DW, Ma Y, Rubin RR, Perreault L, Bray GA, Marrero D, Knowler WC, Barrett-Connor E, Lacoursiere DY; Diabetes Prevention Program Research Group. Depression as a predictor of weight regain among successful weight losers in the diabetes prevention program. Diabetes Care. 2013 Feb;36(2):216-21. doi: 10.2337/dc12-0293. Epub 2012 Sep 21. PMID 23002085
- [Derived] Diabetes Prevention Program Outcomes Study Research Group; Orchard TJ, Temprosa M, Barrett-Connor E, Fowler SE, Goldberg RB, Mather KJ, Marcovina SM, Montez M, Ratner RE, Saudek CD, Sherif H, Watson KE. Long-term effects of the Diabetes Prevention Program interventions on cardiovascular risk factors: a report from the DPP Outcomes Study. Diabet Med. 2013 Jan;30(1):46-55. doi: 10.1111/j.1464-5491.2012.03750.x. PMID 22812594
- [Derived] Perreault L, Pan Q, Mather KJ, Watson KE, Hamman RF, Kahn SE; Diabetes Prevention Program Research Group. Effect of regression from prediabetes to normal glucose regulation on long-term reduction in diabetes risk: results from the Diabetes Prevention Program Outcomes Study. Lancet. 2012 Jun 16;379(9833):2243-51. doi: 10.1016/S0140-6736(12)60525-X. Epub 2012 Jun 9. PMID 22683134
- [Derived] Mather KJ, Christophi CA, Jablonski KA, Knowler WC, Goldberg RB, Kahn SE, Spector T, Dastani Z, Waterworth D, Richards JB, Funahashi T, Pi-Sunyer FX, Pollin TI, Florez JC, Franks PW; Diabetes Prevention Program Research Group. Common variants in genes encoding adiponectin (ADIPOQ) and its receptors (ADIPOR1/2), adiponectin concentrations, and diabetes incidence in the Diabetes Prevention Program. Diabet Med. 2012 Dec;29(12):1579-88. doi: 10.1111/j.1464-5491.2012.03662.x. PMID 22443353
- [Derived] Diabetes Prevention Program Research Group. Long-term safety, tolerability, and weight loss associated with metformin in the Diabetes Prevention Program Outcomes Study. Diabetes Care. 2012 Apr;35(4):731-7. doi: 10.2337/dc11-1299. PMID 22442396
- [Derived] Diabetes Prevention Program Research Group. The 10-year cost-effectiveness of lifestyle intervention or metformin for diabetes prevention: an intent-to-treat analysis of the DPP/DPPOS. Diabetes Care. 2012 Apr;35(4):723-30. doi: 10.2337/dc11-1468. PMID 22442395
- [Derived] Rubin RR, Ma Y, Peyrot M, Marrero DG, Price DW, Barrett-Connor E, Knowler WC; Diabetes Prevention Program Research Group. Antidepressant medicine use and risk of developing diabetes during the diabetes prevention program and diabetes prevention program outcomes study. Diabetes Care. 2010 Dec;33(12):2549-51. doi: 10.2337/dc10-1033. Epub 2010 Aug 30. PMID 20805256
- [Derived] Crandall JP, Polsky S, Howard AA, Perreault L, Bray GA, Barrett-Connor E, Brown-Friday J, Whittington T, Foo S, Ma Y, Edelstein SL; Diabetes Prevention Program Research Group. Alcohol consumption and diabetes risk in the Diabetes Prevention Program. Am J Clin Nutr. 2009 Sep;90(3):595-601. doi: 10.3945/ajcn.2008.27382. Epub 2009 Jul 29. PMID 19640960
- See also: Study website — http://www.dppos.org
- See also: Clinical trials.gov entry for DPP — http://clinicaltrials.gov/ct2/show/NCT00004992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All surviving Diabetes Prevention Program (DPP) participants with consent were invited to enroll into DPPOS throughout the follow-up period. The majority of DPPOS participants were enrolled in 2002-2003.
Pre-assignment Details: DPPOS covers 3 funding phases for the 3 study phases: DPPOS-1 (2002-2008), DPPOS-2 (2009-2014), DPPOS-3 (2015-2021). The groups are defined using the original randomized groups from DPP with recruitment period of 1996-1998.
Groups:
- 1 Original Lifestyle: Boost / Lifestyle, previously Intensive Lifestyle during the DPP
  Group Lifestyle: Quarterly group lifestyle sessions
  Boost Lifestyle: In addition to quarterly group, 2 additional classes per year and an annual 15 minute check-up.
- 2 Original Metformin: Metformin / Lifestyle, previously the metformin treatment group during DPP
  Group Lifestyle: Quarterly group lifestyle sessions
  Metformin: Administered as 850mg twice per day
- 3 Original Placebo: Group Lifestyle, previously placebo treated participants during DPP
  Group Lifestyle: Quarterly group lifestyle sessions
Period: Overall Study
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo
Started | 916 (Includes all enrollees from DPPOS 1-3) | 927 (Includes all enrollees from DPPOS 1-3) | 936 (Includes all enrollees from DPPOS 1-3)
DPPOS Phase 1 Primary | 910 (As reported in the Lancet 2009) | 924 (As reported in the Lancet 2009) | 932 (As reported in the Lancet 2009)
DPPOS Phase 2 Enrolled | 915 (As reported in Lancet Diabetes and Endocrinology 2015) | 926 (As reported in Lancet Diabetes and Endocrinology 2015) | 935 (As reported in Lancet Diabetes and Endocrinology 2015)
DPPOS Phase 2 Primary | 751 (As reported in Lancet Diabetes and Endocrinology 2015) | 772 (As reported in Lancet Diabetes and Endocrinology 2015) | 780 (As reported in Lancet Diabetes and Endocrinology 2015)
DPPOS Phase 3 Enrolled (As of February 2016) | 916 | 927 | 936
Completed | 916 | 927 | 936
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Original Lifestyle: randomized to unmasked Intensive Lifestyle (ILS) during the DPP and offered Intensive Lifestyle Group Session, DPPOS Group Lifestyle plus DPPOS Boost Lifestyle sessions in DPPOS Phase 1 and 2
  DPPOS Group Lifestyle: Quarterly group lifestyle sessions
  DPPOS Boost Lifestyle: In addition to quarterly group, 2 additional classes per year and an annual 15 minute check-up.
  Intensive Lifestyle Group Session: 16 session curriculum in group format. In DPP delivered to ILS as individual sessions
- Total: Total of all reporting groups
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo | Total
Number analyzed (Participants) | 916 | 927 | 936 | 2779
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: An additional 3 participants were enrolled after publication
  years
    number analyzed (Participants) | 915 | 927 | 936 | 2778
    (all) | 54 (11) | 54 (10) | 54 (10) | 54 (10)
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (11.1) | 51.3 (10.1) | 50.7 (10.0) | 51.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 624 | 620 | 645 | 1889
  Male | 292 | 307 | 291 | 890
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 54 | 46 | 55 | 155
  Asian | 44 | 28 | 40 | 112
  Native Hawaiian or Other Pacific Islander | 8 | 1 | 1 | 10
  Black or African American | 173 | 182 | 189 | 544
  White | 596 | 628 | 612 | 1836
  More than one race | 19 | 21 | 19 | 59
  Unknown or Not Reported | 22 | 21 | 20 | 63
Region of Enrollment [Number; unit: participants]
  United States | 916 | 927 | 936 | 2779
BMI [Mean (Standard Deviation); unit: kg/m2] | 33.7 (6.5) | 33.8 (6.5) | 34.0 (6.5) | 33.8 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Development of Diabetes.
Description: Primary outcome for years 2002-2008 defined according to American Diabetes Association criteria (fasting plasma glucose level >= 126 mg/dL [7.0 mmol/L] or 2-hour plasma glucose >= 200 mg/dL [11.1 mmol/L], after a 75 gram oral glucose tolerance test (OGTT), and confirmed with a repeat test).
Time Frame: Outcomes were assessed from 1996-2008 (approximately 12 years including 6 years of DPP).
Measure: Number (95% Confidence Interval); unit: diabetes incidence (cases per 100 person
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo
Number analyzed (Participants) | 916 | 927 | 936
diabetes incidence (cases per 100 person | 5.3 [4.8 to 5.8] | 6.4 [5.9 to 7.1] | 7.8 [7.2 to 8.6]

2. Primary Outcome: Prevalence of Aggregate Microvascular Complication
Description: Aggregate microvascular disease is defined as the average prevalence of 3 components: (1) retinopathy measured by photography (ETDRS of 20 or greater); (2) neuropathy detected by Semmes Weinstein 10 gram monofilament, and (3) nephropathy based on estimated glomerular filtration rate (eGFR by chronic kidney disease (CKD-Epi) equation ) (<45 ml/min, confirmed) and albumin-to-creatinine ratio in spot urine (> 30mg/gm, confirmed).
Time Frame: Outcomes were assessed from 2012-2013 (approximately 2 years).
Population: Number with microvascular outcome data and included in the primary outcome analysis
Measure: Number (95% Confidence Interval); unit: average percentage of participants
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo
Number analyzed (Participants) | 751 | 772 | 780
average percentage of participants | 11.3 [10.1 to 12.7] | 13 [11.7 to 14.5] | 12.4 [11.1 to 13.8]

3. Primary Outcome: Total Cancer Except Non-melanoma Skin Cancer
Description: All primary incident cancers except non-melanoma skin cancer
Time Frame: Outcomes were assessed from 1996-2020 (approximately 24 years).
Reporting Status: Not Posted, anticipated posting 2022-01

4. Primary Outcome: Major Adverse Cardiovascular Events (MACE): Myocardial Infarction (MI), Stroke, or Cardiovascular Death (CVD)
Description: Defined as MI, stroke and CVD death. These outcomes were collected since randomization and adjudicated by an outcomes committee who are blinded to treatment assignment.
Time Frame: Outcomes were assessed from 1996-2025 (approximately 29 years).
Reporting Status: Not Posted, anticipated posting 2025-06

5. Secondary Outcome: Subclinical Atherosclerosis
Description: Measured using coronary artery calcification (CAC).
Time Frame: Outcomes were assessed from 2012-2013 (approximately 2 years).
Population: DPPOS Participants who met eligibility criteria and consented to have CAC measurements - by sex
Measure: Geometric Mean (95% Confidence Interval); unit: CAC geometric mean in AU
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo
Number analyzed (Participants) | 701 | 679 | 681
CAC geometric mean in AU
  Men: number analyzed (Participants) | 468 | 464 | 486
  Men | 70.1 [45.4 to 108.2] | 40.2 [26.1 to 61.9] | 63.7 [41.3 to 98.3]
  Women: number analyzed (Participants) | 213 | 215 | 215
  Women | 6.0 [4.1 to 8.8] | 6.1 [4.2 to 9.0] | 5.3 [3.6 to 7.8]

6. Secondary Outcome: Cognitive Function
Description: Cognitive function defined as a composite measure constructed from tests of memory (English Spanish Verbal Learning Test) and executive function (word fluency and Digit Symbol Substitution Test ).
Time Frame: Outcomes were assessed in visit years starting in 2010, 2012, 2017, 2020.
Reporting Status: Not Posted, anticipated posting 2022-08

7. Secondary Outcome: Short Physical Performance Battery
Description: Physical function is measured using the short physical performance battery (SPPB), which is comprised of measures of 1) time to walk 3-4 meters, 2) balance, i.e., side-by-side stand, semi-tandem stand, and tandem stand, and 3) repeated chair stands.
Time Frame: Outcomes were assessed in visit years starting in 2010, 2012, 2017, 2020.
Reporting Status: Not Posted, anticipated posting 2022-08

8. Secondary Outcome: Frailty
Description: Description: The Cardiovascular Health Study Frailty score is based on 5 frailty characteristics: slow walking speed, low energy expenditure, exhaustion, weak grip strength, and unintentional weight loss.
Time Frame: Outcomes were assessed in visit years starting in 2010, 2012, 2017, 2020.
Reporting Status: Not Posted, anticipated posting 2022-08

9. Secondary Outcome: Mortality
Description: All cause-mortality through clinic reports and National Death Index search
Time Frame: Outcomes were assessed throughout follow-up from 1996 to 2022. National Death Index search conducted in 2019 using early release data as of Dec 2018.
Population: All randomized to DPP were included
Measure: Count of Participants; unit: Participants
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo
Number analyzed (Participants) | 1079 | 1073 | 1082
Participants | 158 | 152 | 143
Statistical Analysis 1: Comparison: 1 Original Lifestyle vs 3 Original Placebo; Test type: Superiority; p = 0.87, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.81 to 1.28]
Statistical Analysis 2: Comparison: 2 Original Metformin vs 3 Original Placebo; Test type: Superiority; p = 0.95, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.79 to 1.25]

ADVERSE EVENTS:
Time Frame: Until data lock of Jan 2014, average of 15 years of follow-up
Arm/Group | 1 Original Lifestyle | 2 Original Metformin | 3 Original Placebo
All-Cause Mortality (participants affected / at risk) | 88/916 | 85/927 | 83/936
Serious Adverse Events (participants affected / at risk) | 472/916 | 482/927 | 492/936
Other Adverse Events (participants affected / at risk) | 234/916 | 274/927 | 257/936
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Original Lifestyle (N=916) | 2 Original Metformin (N=927) | 3 Original Placebo (N=936)
Any SAE Report (General disorders) | 472 (1099) | 482 (1122) | 492 (1103)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 Original Lifestyle (N=916) | 2 Original Metformin (N=927) | 3 Original Placebo (N=936)
Sprains and fractures requiring medical attention (Musculoskeletal and connective tissue disorders) | 234 | 274 | 257

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT00038727/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT00038727/ICF_003.pdf